CLINICAL TRIAL: NCT06522633
Title: Prospective Evaluation of Opioid Withdrawal in Patients With Suspected Opioid-induced Esophageal Dysfunction (OIED)
Brief Title: Esophageal Dysfunction Associated With Opioids: Clinical Response and Manometric Findings After Opioid Discontinuation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Vall Hebron Insitut Recerca (Network)
Responsible Party: Principal Investigator, Elizabeth Barba, Head of Neurogastroenterology and Motility section, Gastroenterology department, Hospital Clinic of Barcelona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HCB/2022/0458
Record Dates: First submitted 2024-06-30; First posted 2024-07-26 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Opioid Use
Keywords: Opioid-Associated Esophageal Dysfunction, dysphagia, esophageal motility
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: In patients under regular treatment with opioids referred to the motility unit for dysphagia, esophageal manometry is performed and if they present an OIED, the morphine is removed and the manometry is repeated to evaluated if OIED was resolved with the suspension of opioid
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- patients under treatment with opioids referred for study of non-obstructive dysphagia for esophageal (Other): In patients with dysphagia referred for esophageal manometry as part of routine clinical practice, if esophageal dysfunction associated with opioid use is diagnosed, such as type III achalasia, esophagogastric junction outflow obstruction, esophageal spasm, or hypercontractile esophagus, the opioid is discontinued and replaced with another analgesic for 7 days. Esophageal manometry is then repeated to determine if the opioid-induced esophageal dysfunction (OIED) has resolved or persists.
  Interventions: Drug: The intervention involves the discontinuation of the opioid.

INTERVENTIONS:
Drug: The intervention involves the discontinuation of the opioid. — Patients with dysphagia and esophageal manometry indicating opioid-induced esophageal dysfunction (OIED) will have the opioid discontinued, and esophageal manometry will be repeated.

SUMMARY:
Background: Opioid-induced esophageal dysfunction is characterized by altered motility of the esophageal body or impaired function of the esophageal sphincters secondary to chronic opioid use. The diagnosis of this condition is made through high-resolution manometry. Following the discontinuation of opioid treatment, most patients experience a clear symptomatic improvement.

Hypothesis: Opioids induce alterations in esophageal motility and esophageal sphincter function that revert after discontinuation of treatment.

Outcome: To demonstrate through high-resolution esophageal manometry that the manometric alterations described in patients with chronic opioid use are secondary to opioid consumption and disappear after discontinuing use.

Methods: In a group of patients with chronic opioid use and diagnosed with a major esophageal motor disorder through high-resolution esophageal manometry, a new high-resolution manometry will be performed after discontinuing opioid treatment for at least 7 days to assess any changes compared to the previous manometry.

The treating physician will be contacted to inform them about the manometry findings and to consider the possibility of discontinuing opioid treatment. Patients will be informed about the association between opioids and esophageal motor disorders and the benefits of discontinuing the medication to evaluate the resolution of symptoms and the observed disorder.

To avoid complications such as withdrawal syndrome or exacerbation of pain due to the reduction of analgesic medication, an alternative medication protocol will be used according to the recommendations of the psychiatry team associated with functional digestive disorders.

Relevance: This project will determine whether the manometric alterations are primary or secondary to opioid treatment. If it is confirmed that they are secondary to the treatment, opioid treatment can be replaced with another analgesic treatment, and esophageal symptoms will improve without the need for more aggressive therapies.

DETAILED DESCRIPTION:
Background and Current State of the Topic Chronic opioid consumption has been increasing significantly in recent years. While the side effects on the small intestine and colon are well-studied and well-established, their effects on the upper gastrointestinal tract are not fully understood, despite patients reporting numerous symptoms such as dysphagia, nausea, or chest pain. Recently, a new entity known as opioid-induced esophageal dysfunction has been described, defined as a motility disorder of the esophageal body or dysfunction of the sphincters in patients with chronic opioid use. Within this entity, the following motor disorders have been primarily observed: outflow tract obstruction, distal esophageal spasm, type III achalasia, and Jackhammer esophagus. However, more studies are needed to determine the prevalence of opioid-induced esophageal dysfunction in chronic opioid users, as well as to understand if opioids can cause other esophageal motor disorders besides those described. Although an association between chronic opioid use and an increase in the incidence of esophageal motor disorders has been demonstrated, there are no prospective studies proving that discontinuation of opioid treatment results in the resolution of the esophageal motor disorder.

Hypothesis During the performance of high-resolution esophageal manometries in our unit, we have observed a higher prevalence of motor disorders in patients who consume opioids. Our hypothesis, based on the available literature, is that most of these disorders can reverse upon discontinuation of opioid treatment without the need for more aggressive therapies. To test this hypothesis, a high-resolution manometry will be performed again after the patient has discontinued opioid treatment for at least 7 days.

Outcomes

Primary Outcome Measure:

Improvement in Esophageal Motility Description: Evaluate the improvement in esophageal motility in chronic opioid users after discontinuation of opioids.

Measurement Tool: High-resolution esophageal manometry (HREM). Unit of Measure: Manometric parameters (e.g., integrated relaxation pressure (IRP) in mmHg).

Secondary Outcome Measure:

Improvement in Dysphagia Severity Description: Assess the improvement in dysphagia severity in chronic opioid users after discontinuation of opioids.

Measurement Tool: Dysphagia Severity Score. Unit of Measure: Dysphagia score (e.g., a numeric scale from 0 to 10).

Description: Evaluate in chronic opioid users with esophageal motor disorders, the improvement in esophageal motility after discontinuation of opioids evaluated by high-resolution esophageal manometry.

Secondary outcome:

Determine if the symptoms that prompted the esophageal motility study disappear with the discontinuation of opioid treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with dysphagia on chronic treatment with opioids referred for study using high-resolution esophageal manometry in our motility laboratory

Exclusion Criteria:

* Those patients who, due to comorbidities, cannot suspend opioid treatment,
* Patients who do not wish to participate,
* Patients who present any symptoms suggestive of withdrawal or who are not able to suspend opioid treatment due to increased pain or discomfort during the seven days prior to the study
* Patients who have received any definitive treatment for the previously diagnosed motor disorder. (pe. Heller myotomy)
* Patients with gastroesophageal junction surgeries (e.g. Nissen type fundoplication)
* Patients with major esophageal endoscopic procedures (e.g. peroral endoscopic myotomy POEM).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Improvement in Esophageal Motility Demonstrate the improvement in esophageal motility in chronic opioid users after discontinuation of opioids. | Baseline (prior to opioid discontinuation) and 7 days post-opioid discontinuation
  Assessment Tool: High-resolution esophageal manometry (HREM). Unit of Measure: Manometric parameters (e.g., integrated relaxation pressure (IRP) in mmHg).
  Prospective multicenter study in patients referred for non-obstructive dysphagia that were on chronic opioid treatment (> 3 months).
  Patients were evaluated during the initial referral and then after 7 days without opioid use.
  In each visit, patients underwent a high-resolution esophageal manometry following the Chicago 4.0 protocol.

SECONDARY OUTCOMES:
Improvement in Dysphagia Severity Demonstrate the improvement in dysphagia severity in chronic opioid users after discontinuation of opioids. | Baseline (prior to opioid discontinuation) and 7 days post-opioid discontinuation
  Change in dysphagia severity
  -Assessment Tool: Dysphagia Severity Score. Unit of Measure: Dysphagia score (numeric scale). Assessment Points: Baseline (during opioid treatment) and after 7 days of opioid discontinuation.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínic of Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Snyder DL, Crowell MD, Horsley-Silva J, Ravi K, Lacy BE, Vela MF. Opioid-Induced Esophageal Dysfunction: Differential Effects of Type and Dose. Am J Gastroenterol. 2019 Sep;114(9):1464-1469. doi: 10.14309/ajg.0000000000000369. PMID 31403963
- [Result] Snyder DL, Vela MF. Impact of opioids on esophageal motility. Neurogastroenterol Motil. 2023 May;35(5):e14587. doi: 10.1111/nmo.14587. Epub 2023 Apr 15. PMID 37060333
- [Result] Kraichely RE, Arora AS, Murray JA. Opiate-induced oesophageal dysmotility. Aliment Pharmacol Ther. 2010 Mar;31(5):601-6. doi: 10.1111/j.1365-2036.2009.04212.x. Epub 2009 Dec 8. PMID 20003176
- [Derived] Ezquerra-Duran A, Alcala-Gonzalez L, Araujo IK, Alcedo J, Serra J, Barba-Orozco E. Prospective Evaluation of Opioid Cessation in Patients With Suspected Opioid-Induced Esophageal Dysfunction. Am J Gastroenterol. 2025 Jan 10;120(6):1400-1404. doi: 10.14309/ajg.0000000000003297. PMID 39791564